CLINICAL TRIAL: NCT00159419
Title: Bisphosphonate Therapy for Osteogenesis Imperfecta
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Linda DiMeglio, MD, MD, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9902-30
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Osteogenesis Imperfecta; Osteoporosis; Paget Disease of Bone
Keywords: Osteogenesis Imperfecta; Fractures; Pediatric; Osteoporosis; Juvenile Pagets
MeSH Terms: conditions — Osteogenesis Imperfecta; Osteoporosis; Osteitis Deformans; Fractures, Bone | interventions — Alendronate; Pamidronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alendronate (Active Comparator): 1 mg/kg po qd rounded to nearest 10 or 20 mg dose
  Interventions: Drug: Alendronate
- Pamidronate (Active Comparator): 3 mg/kg IV q4 months
  Interventions: Drug: Pamidronate

INTERVENTIONS:
Drug: Alendronate
  Other Names: fosamax
  Arms: Alendronate
Drug: Pamidronate
  Arms: Pamidronate

SUMMARY:
The study is designed to evaluate the efficacy and safety of "Bisphosphonate Therapy for Osteogenesis Imperfecta (OI)." We, the researchers at Indiana University School of Medicine, are characterizing the changes effected by oral bisphosphonate therapy and comparing them to a regimen of intravenous bisphosphonate therapy in a group of children with OI and also in children with other disorders that result in low bone mass and fractures.

DETAILED DESCRIPTION:
The study is designed to evaluate the efficacy and safety of "Bisphosphonate Therapy for Osteogenesis Imperfecta (OI)." OI is an inherited disorder of collagen synthesis. Collagen is the major structural protein of the matrix of tendons, skin, and bones. Affected persons have low bone mineral density (and experience multiple fractures and progressive bony deformity). In its most severe form, the disorder is lethal in infancy. We plan to characterize the changes effected by oral bisphosphonate therapy and compare them to a regimen of intravenous bisphosphonate therapy in a group of children with OI.

Additionally, we have begun to treat patients with OI and other conditions of low bone mineralization for age who are not eligible for the standard protocol (too young, history of abdominal pain, etc.) with bisphosphonate. We also plan to screen the parents and siblings of our patients diagnosed with osteogenesis imperfecta, in order to determine if they also have osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OI, as defined by genetic analysis revealing a defect of type I collagen, OR by bone mineral density (BMD) <2.5 standard deviations (SD) for age plus two of the following:

  * Family history of OI
  * Frequent fractures
  * Blue sclerae
  * Multiple wormian bones on skull x-ray
  * Hearing disturbance
  * Dentinogenesis imperfecta
* Age between 3 and 21 years at the start of the study period.
* Children must be able to swallow whole tablets
* Parents of children must be able to understand protocol and give informed consent.

Exclusion Criteria:

* Therapy with bisphosphonates during the past 12 months.
* Other "non-traditional" therapy for OI in the last 6 months, such as growth hormone or anabolic steroids.
* Other chronic diseases besides OI that interfere with bone morphology or gastrointestinal absorption

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 1999-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A DiMeglio, MD, MPH, Principal Investigator — Indiana University School of Medicine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from clinics
Period: Overall Study
Arm/Group | Pamidronate Treatment | Alendronate Treatment
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pamidronate Treatment | Alendronate Treatment | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 8.4 [3.0 to 13.7] | 9.0 [3.8 to 12.7] | 8.7 [3.0 to 13.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density
Description: By Dual-energy x-ray absorptiometry. Results were reported as z-scores as well as as absolute values. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate a better outcome", or similar, as accurate and appropriate.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Pamidronate Treatment | Alendronate
Number analyzed (Participants) | 9 | 9
z-score | -1.3 (2.0) | -1.1 (1.2)

ADVERSE EVENTS:
Groups:
- Pamidronate Treatment: Acute phase reaction with infusion
Arm/Group | Pamidronate Treatment | Alendronate Treatment
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 7/9 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pamidronate Treatment (N=9) | Alendronate Treatment (N=9)
Acute Phase Reaction (General disorders) | 7 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No